CLINICAL TRIAL: NCT01528852
Title: Efficacy of Use of Chlorhexidine to Clean Umbilical Cord of Neonates in First 10 Days for Reduction in Neonatal Mortality and Omphalitis - A Community Based Randomized, Double Masked Controlled Trial in Pemba Tanzania
Brief Title: Chlorhexidine Cordcare for Reduction in Neonatal Mortality and Omphalitis
Acronym: CHX-Pemba
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Annamalai University (Other); Ministry of Health and Social Welfare, Zanzibar (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00003027
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Mortality; Cord Care; Omphalitis
Keywords: neonatal Mortality; chlorhexidine cord care; cord infections; african settings; clinical trials

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CHX Cord application (Experimental): Chlorhexidine cord application for 10 days
  Interventions: Drug: Chlorhexidine 4%
- Control (Active Comparator): Same liquid as intervention without the chlorhexidine used for cord cleaning for 10 days once daily
  Interventions: Other: Control cord cleaning solution
- Dry Cord care (No Intervention): Use current recommended keep cord dry

INTERVENTIONS:
Drug: Chlorhexidine 4% — 4% liquid solution used for cord cleaning once daily for 10 days
  Arms: CHX Cord application
Drug: Chlorhexidine 4% — Chlorhexidine 4% liquid solution used for cord cleaning once daily for 10 days
  Arms: CHX Cord application
Other: Control cord cleaning solution — Mild soapy solution used to clean cord once daily for 10 days
  Arms: Control

SUMMARY:
In a community-based controlled trial among children to evaluate if use of 4% Chlorhexidine cleansing solution on umbilical cord of infants in first 10 days of life results in

* Reduction in neonatal mortality (deaths in first 28 days of life)
* Reduction in umbilical cord infections (defined by moderate or severe redness of the cord) during first 28 days of life
* Reduction in umbilical cord infections (defined by pus formation with any degree of redness) during first 28 days of life.

The double blind part of study uses a control preparation without chlorhexidine (CHX) as control group while in the sub-study dry cord care group is also evaluated as second control. Hypothesis is that CHX group will have lower mortality and umbilical cord infections while control group and dry cord group will be similar as shown in a previous study in Nepal.

DETAILED DESCRIPTION:
Project Goal: The purpose of the trial is to evaluate the efficacy of cord cleansing with Chlorhexidine in the first 10 days of life in reducing neonatal mortality and morbidity. The study would provide a proof of principle for an intervention that could easily be scaled up.

Objectives of formative phase:

* Using TIPS (Trials of Improved Practices) methodology to evaluate the acceptance and impediments if any to practice of using liquid solution for cord cleaning including washing of hands with soap before and after use.
* To compare 3 modes (3 different packaging with application using cotton ball, dropper bottle and squeeze tube) of delivery for cord cleaning in terms of acceptance, ease of use and effectiveness in covering the target area.

Objectives of the main Trial :

Primary Objectives: In a double-blind community-based randomized controlled trial among 24,000 children to evaluate the efficacy of application of 4% Chlorhexidine cleansing solution on umbilical cord of infants in first 10 days of life compared to infants cleansed with a similar control solution without Chlorhexidine for:

* Reduction in neonatal mortality (deaths in first 28 days of life).
* Reduction in umbilical cord infections (defined by moderate or severe redness of the cord) during first 28 days of life.
* Reduction in umbilical cord infections (defined by pus formation with any degree of redness) during first 28 days of life.

Secondary Objectives: In a nested sub-study among 12,000 births (8000 from 24,000 double blind main study and 4000 additional births) randomized to three groups: Chlorhexidine cord care (n=4000), control solution cord care (n=4000) and dry cord care (n=4000):

* To evaluate the sensitivity and specificity of traditionally used "field definitions of omphalitis" based on a combination of signs and symptom in comparison to culture results using state of art sample collection/transport, culture and bacterial identification.
* To evaluate reductions in bacterial colonization rates from a) umbilical cord tip, b) stump and base area in Chlorhexidine and Control Solution groups compared to currently recommended dry cord care.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident of Pemba
* Consenting to participate, infants alive at first contact with MCH/TBA/Hospital staff
* First contact within 48 hours of delivery.

Exclusion Criteria:

* Congenital malformations where application of intervention is not possible
* Very sick child needing hospitalization and ICU care.

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36911 (Actual)
Dates: Start 2011-05-19 (Actual); Primary Completion 2014-09-29 (Actual); Study Completion 2014-09-29 (Actual)

PRIMARY OUTCOMES:
Neonatal Mortality | 28 days after birth

SECONDARY OUTCOMES:
Omphalitis | Birth to 28 days of life
  Using two field based definitions presence of redness or swelling with or without PUS.

CONTACTS AND LOCATIONS:
Locations (1):
- PHL-IDC, Pemba, Zanzibar, Tanzania

REFERENCES:
- [Result] Sazawal S, Dhingra U, Ali SM, Dutta A, Deb S, Ame SM, Mkasha MH, Yadav A, Black RE. Efficacy of chlorhexidine application to umbilical cord on neonatal mortality in Pemba, Tanzania: a community-based randomised controlled trial. Lancet Glob Health. 2016 Nov;4(11):e837-e844. doi: 10.1016/S2214-109X(16)30223-6. Epub 2016 Sep 29. PMID 27693438
- [Derived] Nangia S, Dhingra U, Dhingra P, Dutta A, Menon VP, Black RE, Sazawal S. Effect of 4 % chlorhexidine on cord colonization among hospital and community births in India: a randomized controlled study. BMC Pediatr. 2016 Aug 2;16:121. doi: 10.1186/s12887-016-0625-7. PMID 27484013
- [Derived] Dhingra U, Sazawal S, Dhingra P, Dutta A, Ali SM, Ame SM, Deb S, Suleiman AM, Black RE. Trial of improved practices approach to explore the acceptability and feasibility of different modes of chlorhexidine application for neonatal cord care in Pemba, Tanzania. BMC Pregnancy Childbirth. 2015 Dec 28;15:354. doi: 10.1186/s12884-015-0760-4. PMID 26711437
- [Derived] Dhingra U, Gittelsohn J, Suleiman AM, Suleiman SM, Dutta A, Ali SM, Gupta S, Black RE, Sazawal S. Delivery, immediate newborn and cord care practices in Pemba Tanzania: a qualitative study of community, hospital staff and community level care providers for knowledge, attitudes, belief systems and practices. BMC Pregnancy Childbirth. 2014 May 22;14:173. doi: 10.1186/1471-2393-14-173. PMID 24885689
- See also: Efficacy of chlorhexidine application to umbilical cord on neonatal mortality in Pemba, Tanzania: a community-based randomised controlled trial — https://pubmed.ncbi.nlm.nih.gov/27693438/